CLINICAL TRIAL: NCT04994301
Title: Lung T1 MRI Assessments of Children with CF Initiating Trikafta Therapy
Brief Title: Evaluation of Lung T1-MRI in Pediatric Cystic Fibrosis Patients
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly McBennett, MD, PhD, FACP, Senior Staff Physician, Adult Cystic Fibrosis Center, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20200689
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Transmembrane; Conductance; Regulator
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Oropharyngeal swab for the extraction of bacterial DNA only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with Cystic Fibrosis: Patients (male, female) age 5-11 with confirmed diagnosis of Cystic Fibrosis. These patients will begin clinically prescribed FDA-approved Trikafta therapy.
  Interventions: Diagnostic Test: Lung T1 MRI

INTERVENTIONS:
Diagnostic Test: Lung T1 MRI — Evaluation of lung T1 MRI to Assess Lung Disease

SUMMARY:
In this observational study, the investigators evaluate the sensitivity of T1-MRI to identify lung perfusion changes in pediatric patients with CF (age = 6-11) before and after initiating FDA-approved Trikafta therapy. The investigators compare these Lung T1 MRI assessments (% Normal lung perfusion) to currently best-available assessments of lung function in CF patients (i.e., MBW (LCI( and Spirometry (FEV1 % Predicted).

DETAILED DESCRIPTION:
This is a prospective study with 3 study visits to evaluate the utility of Magnetic Resonance Imaging (MRI) and clinical lung function assessments to detect changes in Cystic Fibrosis (CF) patients before and after administration of the FDA-approved Trikafta therapy. The 3 study visits include:

Visit 1: Before starting Trikafta Visit 2: 3 months from start of Trikafta Visit 3: 6 months from start of Trikafta

Along with the clinical assessments (MBW and Spirometry), all participants will undergo an MRI scan of the lungs to generate quantitative lung T1 maps. The investigators will compare the lung T1 MRI (% Normal Lung Perfusion) to Multiple Breath Washout (LCI) and spirometry (FEV1 % Predicted) as methods to assess lung changes with administration of Trikafta. The investigators will obtain additional clinical assessments from participant's medical records.

This is a multi-site study involving 3 sites.

ELIGIBILITY:
Inclusion Criteria:

• Male or female individuals with a diagnosis of cystic fibrosis and have at least one copy of the F508del mutation.

Exclusion Criteria:

* Subject who cannot hold their breath for up to 15 seconds.
* Subjects who are pregnant.
* Subjects with MRI contraindication (e.g., heart pacemaker, heart defibrillator, metal in within the body.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with cystic fibrosis (CF) who are planning to start Trikafta therapy once approved
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Lung T1-MRI | Visit 1: Before starting Trikafta, Visit 2: 3 months (+/- 15 days) from start of Trikafta, Visit 3: 6 months (+/- 30 days) from start of Trikafta
  Evaluate lung T1-MRI (% Normal Lung Perfusion) to assess lung perfusion changes associated with FDA-approved Trikafta therapy in pediatric cystic fibrosis patients.

SECONDARY OUTCOMES:
Spirometry | Visit 1: Before starting Trikafta, Visit 2: 3 months (+/- 15 days) from start of Trikafta, Visit 3: 6 months (+/- 30 days) from start of Trikafta
  Clinical standard pulmonary function test (FEV1 % Predicted).
Multiple breath washout (MBW) | Visit 1: Before starting Trikafta, Visit 2: 3 months (+/- 15 days) after start of Trikafta, Visit 3: 6 months (+/- 30 days) after start of Trikafta
  Multiple breath washout to assess lung clearance index (LCI) applied per CF clinical standard.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Flask, PhD, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - Riley Hospital for Children, Indianapolis, Indiana
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
Unsure if individual data will need to be presented.